CLINICAL TRIAL: NCT01694394
Title: Prevalence of Sub-Clinical Atrial Fibrillation Using an Implantable Cardiac Monitor in Patient With Cardiovascular Risk Factors (ASSERT-II)
Brief Title: Prevalence of Sub-Clinical Atrial Fibrillation Using an Implantable Cardiac Monitor
Acronym: ASSERT-II
Status: Completed | Type: Observational
Sponsor: Population Health Research Institute (Other)
Collaborators: Abbott Medical Devices (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jeff Healey, Associate Professor, McMaster University, Population Health Research Institute
Other Study IDs: ASSERT-II
Record Dates: First submitted 2012-09-23; First posted 2012-09-27 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; implantable cardiac monitor; left atrial enlargement; CHA2DS2 VASc Score; cardiovascular risk
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be collected for NT-ProBNP and hs-Troponin-T
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cohort: Single arm cohort will receive a St. Jude Medical Implantable Cardiac Monitor (Confirm ICM model 2102) for continuous monitoring over the study follow-up period to determine incidence of sub-clinical atrial fibrillation.
  Interventions: Device: Implantable Cardiac Monitor (Confirm ICM model 2102)

INTERVENTIONS:
Device: Implantable Cardiac Monitor (Confirm ICM model 2102) — Patients who meet the study criteria will be implanted with a St. Jude Medical Confirm Implantable Cardiac Monitor (Confirm ICM) model 2102 or other St. Jude Medical ICM with the same capabilities.
  Other Names: St. Jude Medical Confirm ICM model 2102

SUMMARY:
The primary objective of the study is to determine the rate of detection of sub-clinical atrial fibrillation (≥ 5 minutes)within an average of 12 months following implant of the St. Jude Medical Confirm(R) Implantable Cardiac Monitor in patients with known cardiovascular risk factors and left atrial enlargement, but without prior AF.

DETAILED DESCRIPTION:
Title of Study Prevalence of Sub-Clinical Atrial Fibrillation Using an Implantable Cardiac Monitor in Patients with Cardiovascular Risk Factors (ASSERT-II) Short Title ASSERT-II Study Sponsor Population Health Research Institute (Grant in Aid from St. Jude Medical, Inc.) Principal Investigators Dr. J. Healey, Dr. S. Connolly, Dr. M. Alings Central Coordinating Centre Population Health Research Institute Recruitment and Participating Clinical Sites 250 patients from approximately 30 Sites Phase/Regulatory Status Phase IV - Cohort Study Hypothesis Among elderly patients with cardiovascular risk factors and a left atrial diameter ≥ 4.4 cm, but without prior clinical AF, an implanted continuous ECG monitor (St. Jude Medical Confirm® Implantable Cardiac Monitor) will detect subclinical AF (≥ 5 minutes in duration) in 12% or more of patients during an average follow-up of 12 months.

Study Objectives

Primary Objectives:

1. To determine the rate of detection of sub-clinical atrial AF (≥ 5 minutes) within an average of 12 months following implant of the St. Jude Medical Confirm® Implantable Cardiac Monitor in patients with known cardiovascular risk factors and left atrial enlargement, but without prior AF.

Secondary Objectives

1. To determine if the incidence of sub-clinical AF is higher among patients whose left atrial volume is above the median value observed in this study.
2. To determine the relationship between left atrial volume (continuous variable) and the risk of sub-clinical AF.
3. To evaluate other potential predictors of sub-acute AF in this population including: baseline troponin-T, baseline NT-pro-BNP as well as clinical and other echocardiographic parameters.
4. To develop a preliminary economic analysis to evaluate the potential cost-effectiveness of screening this patient population with an Implantable Cardiac Monitor as a means of preventing stroke.

Study Design Cohort study to determine the prevalence of sub-clinical AF in an elderly population with common cardiovascular risk factors, such as hypertension and diabetes. Patients with echocardiographic evidence of atrial enlargement will be enrolled and have the St. Jude Medical Confirm® Implantable Cardiac Monitor (Confirm® ICM) subcutaneously implanted. To reduce costs, in most cases the implant will be done in conjunction with other planned surgery or heart catheterization.

PHRI: CONFIDENTIAL Final Version 2.0:2012-06-18 Page 4 of 24 Participants/Study Duration Total of 250 participants will be enrolled over 16 months. The last patient enrolled will have 9 months of follow-up, for a total study duration of approximately 25 months. Clinic visits will occur at enrolment and months 3, 6 and 9. A final visit will take place at 18 months of follow-up, or after the last patient enrolled has been followed for 9 months (whichever comes first).

Study Population Patients with known cardiovascular risk factors and left atrial enlargement, with no prior documented AF.

Intervention St. Jude Medical Confirm® Implantable Cardiac Monitor (Confirm® ICM) Enrollment and Follow-up Eligible and consenting patients will be enrolled and have the Confirm® ICM implanted. The implant may take place in conjunction with pre-planned non-cardiac surgery, heart catheterization, or as a stand-alone procedure. Follow-up visits will occur at month 3, 6 and 9. A final visit will take place at 18 months of follow-up, or after the last patient enrolled has been followed for 9 months (whichever comes first).

Assessment of Outcome Events An independent central adjudication committee comprised of arrhythmia experts will evaluate device-detected AF episodes.

Statistical Methodology Determine the incidence of sub-clinical atrial AF (≥ 5 minutes) using the Confirm® ICM.

Date of Protocol June 18, 2012

ELIGIBILITY:
Inclusion Criteria

Patients will be eligible for inclusion if they meet both of the following:

1. Age ≥ 65, plus:

   * CHA2DS2-VASc score ≥ 2 Or
   * Obstructive sleep apnea (documented by polysomnography, ambulatory oximetry, positive Berlin Questionnaire or requiring the use of CPAP/BiPAP) Or
   * BMI > 30
2. Echocardiographic or biochemical evidence of increased risk of AF:

   * Left atrial enlargement on a clinical echocardiography at any time prior to enrollment ( defined as LA volume ≥ 58 ml or LA diameter of ≥ 4.4 cm) Or
   * Serum NT-ProBNP ≥ 290 pg/mL Exclusion Criteria

1. Previously documented history of atrial fibrillation or atrial flutter 2. Current chronic treatment with oral anticoagulation (i.e. those on peri-operative prophylaxis would be eligible) 3. Patient with implanted pacemaker or defibrillator with an atrial lead 4. Definitive plan for cardiac surgery in the next 6 months (patients who are having coronary angiography with a possibility of cardiac surgery are still eligible)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients at increased risk of atrial fibrillation and cardiovascular events but without prior history of atrial fibrillation or implanted pacemaker or defibrillator
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2012-12; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
First atrial fibrillation episode at least 5 minutes in duration | over maximum follow-up of 18 months
  incidence of atrial fibrillation detected by continuous monitoring by an implantable cardiac monitor

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Healey, M.D., Principal Investigator — Population Health Research Institute; Stuart Connolly, M.D., Principal Investigator — Population Health Research Institute; Marco Alings, M.D., Principal Investigator — Working group Cardiovascular research Netherlands
Locations (19):
- Canada (13):
  - University of Calgary, Calgary, Alberta
  - St. Boniface Hospital, Winnepeg, Manitoba
  - Queen Elizabeth-II Heather Sciences Center, Halifax, Nova Scotia
  - Health Sciences North, Greater Sudbury, Ontario
  - Hamilton Health Sciences - Electrophysiology Clinic, Hamilton, Ontario
  - Hamilton Health Sciences - Interventional Cardiology, Hamilton, Ontario
  - Hamilton Health Sciences - Perioperative Ischemia Research Group, Hamilton, Ontario
  - London Health Sciences Center University Hospital, London, Ontario
  - Southlake Regional HealthCare, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Hopital Laval), Sainte-Foy, Quebec
- Netherlands (6):
  - Academisch Medisch Centrum (AMC) Amsterdam, Amsterdam
  - Amphia Hospital, Breda
  - Nij Smellinge, Drachten
  - Groene Hart Ziekenhuis Gouda, Gouda
  - Diakonessenhuis Leiden, Leiden
  - Ikazia Hospital, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Healey JS, Alings M, Ha A, Leong-Sit P, Birnie DH, de Graaf JJ, Freericks M, Verma A, Wang J, Leong D, Dokainish H, Philippon F, Barake W, McIntyre WF, Simek K, Hill MD, Mehta SR, Carlson M, Smeele F, Pandey AS, Connolly SJ; ASSERT-II Investigators. Subclinical Atrial Fibrillation in Older Patients. Circulation. 2017 Oct 3;136(14):1276-1283. doi: 10.1161/CIRCULATIONAHA.117.028845. Epub 2017 Aug 4. PMID 28778946